CLINICAL TRIAL: NCT01900028
Title: A Non-randomised, Open-label, Sequential, Three-part, Phase I Study to Assess the Effect of Itraconazole (a CYP3A4 Inhibitor) on the Pharmacokinetics of Olaparib Following Oral Dosing of a Tablet Formulation, and to Provide Data on the Effect of Olaparib on QT Interval Following Oral Dosing of a Tablet Formulation to Patients With Advanced Solid Tumours
Brief Title: To Assess the Effect of Itraconazole (a CYP3A4 Inhibitor) on the Pharmacokinetics of Olaparib, and the Effect of Olaparib on QT Interval Following Oral Dosing of a Tablet Formulation to Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: D0816C00007; 2013-001892-18 (EudraCT Number)
Record Dates: First submitted 2013-07-12; First posted 2013-07-16 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Solid Tumours
Keywords: oncology,; cancer,; tumour,; anticancer drug,; pharmacokinetics,; olaparib,itraconazole,; neoplasm,; QT interval
MeSH Terms: conditions — Neoplasms | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Olaparib alone, olaparib+itraconozole (Experimental): Sequential treatments of olaparib alone followed by olaparib+itraconazole, with a washout period in between.
  Interventions: Procedure: Pharmacokinetic sampling; Drug: Olaparib tablet dosing; Drug: Itraconazole

INTERVENTIONS:
Procedure: Pharmacokinetic sampling — Blood samples taken pre and post dosing with olaparib+/- itraconazole
Drug: Olaparib tablet dosing — Olaparib tablets: Part A 100mg od, days 1 and 9 only. Part B 10x300mg doses over 5 days (300mg bd).
Drug: Itraconazole — Itraconazole 200mg od Part A days 5 to 11 only

SUMMARY:
This is a 3-part study in patients with advanced solid tumours: Part A will assess the effect of itraconazole on the PK parameters of olaparib and will determine the effect of olaparib on the QT interval following single oral dosing; Part B will determine the effect of olaparib on the QT Interval following multiple oral dosing; Part C will allow patients continued access to olaparib after the PK and QT phases and will provide for additional safety data collection. A total of 48 patients are planned to be enrolled; at least 42 evaluable patients will be required to complete the study. Patients will participate as a single cohort in all parts of the study.

ELIGIBILITY:
Inclusion criteria:-

For inclusion in the study, patients should fulfil the following criteria:

1. Provision of written informed consent prior to any study-specific procedures.
2. Patients aged greater than or equal to 18 years.
3. Histologically or, where appropriate, cytologically confirmed malignant solid tumour refractory or resistant to standard therapy or for which no suitable effective standard therapy exists.
4. Patients must have normal organ and bone marrow function measured within 28 days prior to administration of investigational product (IP) as defined below: Haemoglobin (Hb) greater than or equal to 10.0 g/dL, with no blood transfusions in the previous 28 days. Absolute neutrophil count (ANC) greater than or equal to 1.5 x 109/L. White blood cells (WBC) greater than 3 x 109/L. Platelet count greater than or equal to 100 x 109/L. Total bilirubin less than or equal to 1.5 x institutional upper limit of normal (ULN) (except in the case of Gilbert's disease). Aspartate aminotransferase (AST), alanine aminotransferase (ALT) less than or equal to 2.5 x institutional ULN unless liver metastases are present in which case it must be less than or equal to 5x ULN. Serum creatinine less than or equal to 1.5 x institutional ULN. Serum potassium, sodium, magnesium and calcium within the institutional normal range.
5. Calculated serum creatinine clearance greater than 50 mL/min (using Cockroft-Gault formula or by 24 hour urine collection).
6. Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2. 7. Patients must have a life expectancy of greater than or equal to 16 weeks.

8. Evidence of non-childbearing status for women of childbearing potential, or post-menopausal status: negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on Day 1 of Part A. Post-menopausal is defined as: Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments. Luteinising hormone and follicle stimulating hormone levels in the post-menopausal range for women under 50 years of age. Radiation-induced oophorectomy with last menses greater than1 year ago. Chemotherapy-induced menopause with greater than1 year interval since last menses. Surgical sterilisation (bilateral oophorectomy or hysterectomy).

9. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.

10. Patients must be on a stable concomitant medication regimen (with the exception of electrolyte supplements), defined as no changes in medication or in dose within the 2 weeks prior to start of olaparib dosing, except for bisphosphonates, denosumab, and corticosteroids, which should be at a stable dose for at least 4 weeks prior to the start of olaparib dosing.

Exclusion criteria:-

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

1. Involvement in the planning and/or conduct of the study (applies to AstraZeneca staff, its agents, and/or staff at the study site).
2. Previous enrolment in the present study.
3. Participation in another clinical study with an IP during the last 14 days (or a longer period depending on the defined characteristics of the agents used).
4. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 2 weeks prior to study treatment (or a longer period depending on the defined characteristics of the agents used). The patient can receive a stable dose of bisphosphonates or denosumab for bone metastases, before and during the study, as long as these were started at least 4 weeks prior to treatment.
5. Patients who have received or are receiving inhibitors or inducers of CYP3A4.
6. Toxicities (greater than or equal to CTCAE Grade 2) caused by previous cancer therapy, excluding alopecia.
7. Any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days of the first administration of the IP until the end of Part A.
8. Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. Patients with asymptomatic brain metastases or with symptomatic but stable brain metastases can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment.
9. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
10. Patients unable to fast for up to 14 hours.
11. Patients considered a poor medical risk due to a serious uncontrolled medical disorder, non malignant systemic disease, uncontrolled seizures, or active uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive bilateral interstitial lung disease on high resolution computer tomography (HRCT) scan, or any psychiatric disorder that prohibits obtaining informed consent.
12. Patients with a history of poorly controlled hypertension with resting blood pressure (BP) greater than150/100 mm Hg in the presence or absence of a stable regimen of hypertensive therapy. Measurements will be made after the patient has been resting supine for a minimum of 5 minutes. Two or more readings should be taken at 2 minute intervals and averaged. If the first 2 diastolic readings differ by more than 5 mm Hg, an additional reading should be obtained and averaged.
13. Patients with a history of heart failure, or left ventricular dysfunction, and patients who require calcium channel blockers.
14. Patients who have gastric, gastro-oesophageal or oesophageal cancer.
15. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders or significant gastrointestinal resection likely to interfere with the absorption of Olaparib.
16. Breastfeeding women.
17. Immunocompromised patients, eg, patients who are known to be serologically positive for human immunodeficiency virus (HIV).
18. Patients with known active hepatic disease (ie, hepatitis B or C).
19. Patients with a known hypersensitivity to itraconazole or any of the excipients of the product.
20. Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
21. Mean QTc with Fridericia's correction (QTcF) greater than 470 ms in screening ECG or history of familial long QT syndrome:

    A marked baseline prolongation of QT/QTc interval (eg, repeated demonstration of a QTc interval greater than 470 ms).

    A history of additional risk factors for Torsade de pointes (eg, heart failure, hypokalaemia, family history of long QT syndrome).
22. The use of concomitant medications that prolong the QT/QTc interval.
23. Concomitant medication contraindicated for use with itraconazole (including, but not limited to): cisapride, oral midazolam, nisoldipine, pimozide, quinidine, dofetilide, triazolam, levacetylmethadol (levomethadyl), 3-hydroxy-3-methyl-glutaryl coenzyme A (HMG-CoA)-reductase inhibitors metabolized by CYP3A4, such as lovastatin and simvastatin, ergot alkaloids metabolized by CYP3A4, such as dihydroergotamine, ergometrine (ergonovine), ergotamine and methylergometrine (methylergonovine).
24. Clinical judgment by the investigator that the patient should not participate in the study

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of olaparib by assessment of maximum plasma olaparib concentration (Cmax) | Blood samples are collected on Day 1& Day 9 at pre-dose, 0.25 , 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post olaparib dose Part A. Part B:Day 5 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose
  Rate and extent of absorption of olaparib following single (Part A) and multiple (Part B) oral doses of olaparib tablet formulation by assessment of maximum plasma olaparib concentration (Cmax)
Pharmacokinetics of olaparib by assessment of area under the plasma concentration time curve from zero to infinity (AUC) | Blood samples are collected on Day 1& Day 9 at pre-dose, 0.25 , 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post olaparib dose Part A. Part B:Day 5 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose
  Rate and extent of absorption of olaparib following single (Part A) and multiple (Part B) oral doses of olaparib tablet formulation by assessment of area under the plasma concentration time curve from zero to infinity (AUC)
Pharmacokinetics of olaparib by assessment of area under the plasma concentration time curve from zero to the last measurable time point, AUC0-t, if AUC is not adequately estimable). | Blood samples are collected on Day 1& Day 9 at pre-dose, 0.25 , 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post olaparib dose Part A. Part B:Day 5 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose
  Rate and extent of absorption of olaparib following single (Part A) and multiple (Part B) oral doses of olaparib tablet formulation by assessment of area under the plasma concentration time curve from zero to the last measurable time point, (AUC0-t)

SECONDARY OUTCOMES:
Pharmacokinetics of olaparib by assessment of time to reach maximum plasma concentration for olaparib (tmax) | PK samples taken on Day 1 & Day 9 at pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, & 72 hours post dose (Part A). And in Part B, Day 5 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose
  Rate and extent of absorption of olaparib following following single (Part A) and multiple (Part B) oral doses of olaparib tablet formulation by assessment of time to reach maximum plasma concentration for olaparib (tmax)
Pharmacokinetics of olaparib by assessment of area under the plasma concentration time curve from zero to the last measurable time point (AUC0-τ) | PK samples taken on Day 1 & Day 9 at pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, & 72 hours post dose (Part A). And in Part B, Day 5 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose
  Rate and extent of absorption of olaparib following following single (Part A) and multiple (Part B) oral doses of olaparib tablet formulation by assessment of area under the plasma concentration time curve from zero to the last measurable time point (AUC0-τ)
Pharmacokinetics of olaparib by assessment of time olaparib apparent clearance (CL/F) | PK samples taken on Day 1 & Day 9 at pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, & 72 hours post dose (Part A). And in Part B, Day 5 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose
  Rate and extent of absorption of olaparib following following single (Part A) and multiple (Part B) oral doses of olaparib tablet formulation by assessment of time olaparib apparent clearance (CL/F)
Pharmacokinetics of olaparib by assessment of olaparib apparent volume of distribution (Vz/F) | PK samples taken on Day 1 & Day 9 at pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, & 72 hours post dose (Part A). And in Part B, Day 5 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose
  Rate and extent of absorption of olaparib following following single (Part A) and multiple (Part B) oral doses of olaparib tablet formulation by assessment of olaparib apparent volume of distribution (Vz/F)
Pharmacokinetics of olaparib by assessment of olaparib terminal half-life (t1/2). | PK samples taken on Day 1 & Day 9 at pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, & 72 hours post dose (Part A). And in Part B, Day 5 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose
  Rate and extent of absorption of olaparib following following single (Part A) and multiple (Part B) oral doses of olaparib tablet formulation by assessment of olaparib terminal half-life (t1/2).
Pharmacokinetics of itraconazole by assessment of maximum plasma itraconazole concentration (Cmax) | PK samples taken on Day 1 & Day 9 at pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, & 72 hours post dose (Part A). And in Part B, Day 5 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose
  Rate and extent of absorption of itraconazole by assessment of maximum plasma itraconazole concentration (Cmax).
Pharmacokinetics of itraconazole by assessment of area under the plasma concentration time curve from zero to the last measurable time point (AUC0-τ), | PK samples taken on Day 1 & Day 9 at pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, & 72 hours post dose (Part A). And in Part B, Day 5 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose
  Rate and extent of absorption of itraconazole by assessment of area under the plasma concentration time curve from zero to the last measurable time point (AUC0-τ)
Pharmacokinetics of itraconazole by assessment of time to reach maximum plasma concentration for itraconazole (tmax) | PK samples taken on Day 1 & Day 9 at pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, & 72 hours post dose (Part A). And in Part B, Day 5 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose
  Rate and extent of absorption of itraconazole by assessment of time to reach maximum plasma concentration for itraconazole (tmax)
Pharmacokinetics of itraconazole by assessment of itraconazole apparent clearance (CL/F) | PK samples taken on Day 1 & Day 9 at pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, & 72 hours post dose (Part A). And in Part B, Day 5 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose
  Rate and extent of absorption of itraconazole by assessment of itraconazole apparent clearance (CL/F)
Pharmacokinetics of hydroxy-itraconazole by assessment of maximum plasma hydroxyl -itraconazole concentration (Cmax). | PK samples taken on Day 1 & Day 9 at pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, & 72 hours post dose (Part A). And in Part B, Day 5 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose
  Rate and extent of absorption of hydroxyl -itraconazole by assessment of maximum plasma hydroxyl -itraconazole concentration (Cmax).
Pharmacokinetics of hydroxy-itraconazole by assessment of hydroxy-itraconazole apparent clearance (CL/F) | PK samples taken on Day 1 & Day 9 at pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, & 72 hours post dose (Part A). And in Part B, Day 5 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose
  Rate and extent of absorption of hydroxy-itraconazole by assessment of hydroxy-itraconazole apparent clearance (CL/F)
Pharmacokinetics of hydroxy-itraconazole by assessment of time to reach maximum plasma concentration for hydroxyl-itraconazole (tmax) | PK samples taken on Day 1 & Day 9 at pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, & 72 hours post dose (Part A). And in Part B, Day 5 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose
  Rate and extent of absorption of hydroxyl -itraconazole by assessment time to reach maximum plasma concentration for hydroxyl-itraconazole (tmax)
Pharmacokinetics of hydroxy-itraconazole by assessment of the area under the plasma concentration time curve from zero to the last measurable time point (AUC0-τ) | PK samples taken on Day 1 & Day 9 at pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, & 72 hours post dose (Part A). And in Part B, Day 5 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post dose
  Rate and extent of absorption of hydroxyl -itraconazole by assessment of area under the plasma concentration time curve from zero to the last measurable time point (AUC0-τ)
Assessment of Electrocardiogram (ECG) intervals (including QT and QTc interval) | Digital ECGs recorded Day -1, Day 1 & 9 of Part A: pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, & 24 hours post olaparib dose. In Part B, Day -1, Day 5: pre-dose, 1, 1.5, 2, 3, 4, 6, 8, &12 hours post dose.
  Assessment of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle (the QT interval), uncorrected and corrected for heart rate (QTc) following single (Part A) and multiple (Part B) oral doses of olaparib tablet formulation.
Safety monitoring of olaparib by collection of adverse events | From baseline until 30 days after last dose of olaparib, assessed up to 8 months
  Assessment of adverse events (AEs), graded by CTCAE (v4.0): Adverse events (AEs) will be collected from the time of signed informed consent throughout the treatment period in Part A and Part B up to and including the 30-day follow-up period. In Part C, AEs will be collected until 12 months after the last patient entered Part C, and including the 30 day follow-up period for any patients who discontinue
Safety monitoring of olaparib by collection of physical examination | From baseline until 30 days after last dose of olaparib, assessed up to 8 months
  These will occur at screening, on the day before dosing in each treatment period and 30 days after last dose in Parts A and B. In Part C, will be assessed weekly for a 28-day period followed by every 4 weeks up to 12 months after the last patient enters Part C and at treatment discontinuation. All will be assessed 30 days after last dose.
Safety monitoring of olaparib by collection of vital signs | From baseline until 30 days after last dose of olaparib, assessed up to 8 months
  Assessment of vital signs (including BP and pulse). These will occur at screening, on the day before dosing in each treatment period and 30 days after last dose in Parts A and B. In Part C, all except ECG will be assessed weekly for a 28-day period followed by every 4 weeks up to 12 months after the last patient enters Part C and at treatment discontinuation. All will be assessed 30 days after last dose.
Safety monitoring of olaparib by collection of clinical laboratory results | From baseline until 30 days after last dose of olaparib, assessed up to 8 months
  Assessment of laboratory parameters (clinical chemistry, hematology, and urinalysis) : These will occur at screening, on the day before dosing in each treatment period and 30 days after last dose in Parts A and B. In Part C, all except ECG will be assessed weekly for a 28-day period followed by every 4 weeks up to 12 months after the last patient enters Part C and at treatment discontinuation. All will be assessed 30 days after last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Anitra Fielding, Study Director — AstraZeneca Senior Research Physician; Ruth Plummer, Prof, Principal Investigator — Northern Centre for Cancer Care, Newcastle Upon Tyne
Locations (11):
- Belgium (3):
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
- Denmark (2):
  - Research Site, Copenhagen
  - Research site, Herlev
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Maastricht
  - Research Site, Nijmegen
- United Kingdom (3):
  - Research Site, London
  - Research Site, Newcastle
  - Research Site, Sutton

REFERENCES:
- [Derived] Dirix L, Swaisland H, Verheul HM, Rottey S, Leunen K, Jerusalem G, Rolfo C, Nielsen D, Molife LR, Kristeleit R, Vos-Geelen J, Mau-Sorensen M, Soetekouw P, van Herpen C, Fielding A, So K, Bannister W, Plummer R. Effect of Itraconazole and Rifampin on the Pharmacokinetics of Olaparib in Patients With Advanced Solid Tumors: Results of Two Phase I Open-label Studies. Clin Ther. 2016 Oct;38(10):2286-2299. doi: 10.1016/j.clinthera.2016.08.010. Epub 2016 Oct 10. PMID 27745744
- See also: D0816C00007_Study_Synopsis_Redacted.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1826&filename=D0816C00007_Study_Synopsis_Redacted.pdf